CLINICAL TRIAL: NCT06935097
Title: Mediterranean Diet Intervention Among Men at LBJ Hospital With Prostate Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-0331; NCI-2025-02780 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention with Mediterranean Diet (Experimental): Twenty-five (25) self-identified Black and/or Hispanic men with newly diagnosed (within 6 months) localized PCa or who have been managed on active surveillance for less than 5 years will be enrolled along with their spouses (if applicable).
  Interventions: Behavioral: Mediterranean diet-based Intervention

INTERVENTIONS:
Behavioral: Mediterranean diet-based Intervention — Through existing collaboration with the Harris Health system's innovative food pharmacy, participants will be provided fresh fruit, vegetables and other foods every other week during the study.
  Participants will receive olive oil and walnuts during the 8 week intervention (consistent with the PREDIMED6 intervention) to supplement their (and their families') diet during the 8-week intervention (while personalized education about diet, food choices and preparation is still occurring).

SUMMARY:
This study, we will build upon our prior work and test the feasibility of a Mediterranean diet intervention for medically underserved men with prostate cancer seen at LBJ Hospital, a large safety net facility in Harris County, TX.

DETAILED DESCRIPTION:
Primary Objectives:

To determine the feasibility of a Mediterranean diet-based intervention adapted for underrepresented minority men with prostate cancer, defined based on the following process measures68:

* Enrollment (completion of 25 patient accrual within 2 years)
* Retention (completion of the study through the 6-month time point, with ≥80% defined as successful)
* Adherence (the percentage of completed study sessions and clinic visits, with ≥70% considered successful).

Secondary Objectives:

To determine changes due to the Mediterranean diet intervention in the following measures:

* Mediterranean diet score (define using MEPA I calculated using VioScreen data)
* Weight/BMI
* QoL (EQ-5D-5L)
* Physical activity (IPAS)
* Non-invasive biomarkers
* Gut microbiome
* Metabolomics

To determine fidelity of intervention,62 including a description of patient comprehension, cognitive skills and perceived ability to change diet during the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate that is localized based on metastatic workup ordered by the treating physician (which may include CT scan, bone scan, MRI and/or other imaging). Note that metastatic workup is not required for enrollment.
* Diagnosis within 12 months prior to enrollment OR
* Currently managed on active surveillance, with initial biopsy being <5 years from date of enrollment
* Self-identified Hispanic and/or Black/African American
* Patient at LBJ Hospital

Exclusion Criteria:

* Special dietary requirements such that patient is unwilling to attempt dietary change
* Unwillingness to participate in study activities
* Inability to keep appointments
* Food allergy prohibitive of a Mediterranean diet, i.e. nuts allergy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males
Enrollment: 25 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Justin Gregg, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Lyndon B Johnson Hospital, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org